CLINICAL TRIAL: NCT03477994
Title: Efficacy of Dexmedetomidine Versus Clonidine to Control Delirium in Patients Undergoing Coronary Artery Bypass Grafting
Brief Title: Efficacy of Dexmedetomidine Versus Clonidine to Control Delirium in Patients Undergoing CABG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hoda Shokri, Hoda Shokri, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FMASU R 16
Record Dates: First submitted 2018-03-20; First posted 2018-03-27 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Delirium on Emergence
Keywords: dexmedetomidine, clonidine, postoperative, CABG
MeSH Terms: conditions — Emergence Delirium | interventions — Dexmedetomidine; Clonidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dexmedetomidine group (Active Comparator): Upon arrival to ICU, in the dexmedetomidine group, patients will receive an infusion of 0.5-0.7 μg/kg/h then 1.4 μg/kg/h if Richmond assessment sedation score from +1 to +4
  +4 Combative ,+3 Very agitated ,+2 Agitated,+1 Restless, 0 Alert and calm, -1 Drowsy , -2 Light sedation, -3 Moderate sedation, -4 Deep sedation, -5 Unarrousable Taking into consideration if the heart rate less than 60 per minute or persistent hypotension reduce infusion rate by 0.2 μg/kg/h. Once the patient will be extubated, wean the infusion by 0.1μg/kg/h till reaching 0.2μg/kg/h. Slow the weaning rate if evidence of withdrawal reactions as agitation or hypertension occur.
  Interventions: Drug: Dexmedetomidine
- clonidine group (Sham Comparator): In clonidine group, the patients will receive 0.5μg/kg then 0.1-0.2 μg/kg/h if Richmond assessment sedation score from +1 to +4 Five ampoules of clonidine(750 μg) will be drawn up and diluted in 45ml of normal saline.
  Interventions: Drug: Clonidine

INTERVENTIONS:
Drug: Dexmedetomidine — an infusion of 0.5-0.7 μg/kg/h then 1.4 μg/kg/h if Richmond assessment sedation score from +1 to +4 ,if the heart rate less than 60 per minute or persistent hypotension reduce infusion rate by 0.2 μg/kg/h.
  Other Names: demedetomidine hydrochloride
  Arms: dexmedetomidine group
Drug: Clonidine — an infusion of 0.5μg/kg then 0.1-0.2 μg/kg/h if Richmond assessment sedation score from +1 to +4.
  Other Names: clonidine hydrochloride
  Arms: clonidine group

SUMMARY:
This prospective, randomised, double blinded, controlled clinical trial will be conducted in 147 patients between 60 yr and 70 yr , ASA physical status II and III, undergoing CABG. Patients will be randomly allocated to either dexmedetomidine or clonidine (control) groups .Upon arrival to ICU, in the dexmedetomidine group, patients will receive an infusion of 0.5-0.7 μg/kg/h then 1.4 μg/kg/h if Richmond assessment sedation score from +1 to +4

Taking into consideration if the heart rate less than 60 per minute or persistent hypotension reduce infusion rate by 0.2 μg/kg/h.

Once the patient will be extubated, wean the infusion by 0.1μg/kg/h till reaching 0.2μg/kg/h. Slow the weaning rate if evidence of withdrawal reactions as agitation or hypertension occur. In clonidine group, the patients will receive 0.5μg/kg then 0.1-0.2 μg/kg/h.Primary end point of the study is the incidence of delirium.The secondary endpoints will be the the duration of extubation, the length of ICU stay, need for inotropic support or vasopressors, hospital stay , mean arterial blood pressure and heart rate , hospital mortality rate , all additional sedatives including overall doses of morphine and haloperidol the incidence of adverse events as bradycardia

DETAILED DESCRIPTION:
After Ethics committee approval, and a written informed consent will be taken from every patient, . Patients with a history of mental illness, severe dementia, delirium or undergoing emergency procedures will be excluded.

Anesthesia management will be standardized to minimize any effect of anesthetic type on neurological outcomes. Premedication with midazolam will be limited to a maximum of 0.05 mg/kg.

Anesthesia will be induced with 12 μg/kg fentanyl, 5-7mg/kg thiopental sodium, and 0.15 mg/kg pancuronium and maintained with 1% to 2.0% isoflurane. The heart rate and blood pressure will be maintained within 20% of the baseline values. Anticoagulation will be achieved with heparin to maintain an activated clotting time above 480 s.The CPB circuit will be primed with 1.8 l lactated Ringer's solution and 50 ml of 20% mannitol. Management of CPB will include systemic temperature drift to 32 C, targeted mean perfusion pressure between 60 and 80 mmHg, and pump flow rates of 2.2 l/min/m2 . Myocardial protection will be achieved with antegrade cold blood cardioplegia. A 32-μ m filter (Avecor Affinity, USA)will be used in the arterial perfusion line. Before separation from CPB, patients will be rewarmed to 36 to 37C. After separation from CPB, heparin will be neutralized with protamine sulfate, 1 mg/100 U heparin, to reach an activated clotting time within 10% of baseline.All patients will be transferred to ICU after surgery. Patients will be randomly allocated to either dexmedetomidine or clonidine (control) groups according to a computer-generated randomization code, with allocation ratio 1:1 .Opaque sealed envelopes will be done according to the randomization schedule and opened by a physician not involved in the study . Upon arrival to ICU, in the dexmedetomidine group, patients will receive an infusion of 0.5-0.7 μg/kg/h then 1.4 μg/kg/h if Richmond assessment sedation score from +1 to +4

+4 Combative ,+3 Very agitated ,+2 Agitated,+1 Restless, 0 Alert and calm, -1 Drowsy , -2 Light sedation, -3 Moderate sedation, -4 Deep sedation, -5 Unarrousable A four millilitres vial of dexmedetomidine ( 100 micrograms per ml)will be drawn up and diluted in 46 ml of normal saline.The infusion of dexmedetomidine will be continued for a maximum period of 24 h. Taking into consideration if the heart rate less than 60 per minute or persistent hypotension reduce infusion rate by 0.2 μg/kg/h.Dexmedetomidine infusion will not be discontinued before extubation. Once the patient will be extubated, wean the infusion by 0.1μg/kg/h till reaching 0.2μg/kg/h. Slow the weaning rate if evidence of withdrawal reactions as agitation or hypertension occur. In clonidine group, the patients will receive 0.5μg/kg then 0.1-0.2 μg/kg/h.

Five ampoules of clonidine(750 μg) was drawn up and diluted in 45ml of normal saline.

Opioids were titrated to reach pain score 3 out of 10. Pain will be assessed using a standard 10-cm visual analog scale (0, no pain; 10, worst and unbearable pain). Patients received 2 mg morphine as rescue analgesic.

Primary end point of the study is the incidence of delirium, which is defined as a disturbed level of consciousness that develops over a period of hours or days and fluctuates over time.

Delirium will be assessed preoperatively (baseline)and postoperatively, in ICU every 2 hours using the confusion assessment method (CAM) for ICU.(7) When patients are discharged from ICU to the ward, delirium will be assessed using CAM every 8 hours for the next 5 days. The CAM-ICU is used for both ventilated and extubated patients. It included a fourstep algorithm : (1) an acute onset of changes or fluctuations in the course of mental status, (2)inattention, (3) disorganized thinking, and (4) an altered level of consciousness. Patients are delirious if both (1) and (2) were found inanition to either feature (3)or (4). Patients are stated either CAM positive (delirium present) or CAM negative (delirium absent). Incidence of delirium was confirmed by the psychiatry consultant. The onset and duration of delirium will be also recorded. The CAM-ICU and CAM testers were involved in the study . IV haloperidol(2.5-5 mg PRN), will be used as a first-line treatment in delirious patients, a regular dose 1 mg ads until symptoms resolve.

The secondary endpoints will be the the duration of extubation, the length of ICU stay, need for inotropic support or vasopressors, hospital stay , mean arterial blood pressure and heart rate , hospital mortality rate , all additional sedatives including overall doses of morphine and haloperidol, finally the incidence of adverse events as bradycardia, heart block , the need for pacemaker , nausea and vomiting will be recorded as well.

ELIGIBILITY:
Inclusion Criteria:

60-70 yrs age ASA II, III Scheduled for CABG -

Exclusion Criteria:

History of mental illness Delirium or dementia patient refusal to participate Emergency procedures Any contraindications to study drugs

-

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
the incidence of delirium | every 4 hours in first day in ICU then every 8h for the next day, after discharge from ICU to the ward it will be checked every 8h for 5 days
  disturbed level of consciousness that develops over a period of hours or days and fluctuates over time.

SECONDARY OUTCOMES:
length of ICU stay | 2 days
  time to stay in ICU discharge to the ward

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Shoeb, professor, Study Chair — Ain Shams University
Locations (1):
- Ain Shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
IPD including protocol will be shared
Supporting Information: Study Protocol, SAP, ICF
Time Frame: about one year
Access Criteria: prevention of delirium post cardiac surgery